CLINICAL TRIAL: NCT03790956
Title: Safety and Efficacy of a Silk Protein Microparticle-based Filler for Injection Augmentation in Treating Unilateral Vocal Fold Paralysis
Brief Title: Silk Protein Microparticle-based Filler for Injection Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Sofregen Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Johns, Professor, Otolaryngology-Head and Neck Surgery; Director, USC Voice Center, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-18-05229
Record Dates: First submitted 2018-11-25; First posted 2019-01-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Vocal Cord Paralysis Unilateral; Dysphonia; Dysphagia, Oropharyngeal
Keywords: vocal fold paralysis; glottal insufficiency; vocal fold injection; augmentation; medialization; laryngoplasty; silk
MeSH Terms: conditions — Vocal Cord Paralysis; Dysphonia; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Single vocal fold injection of study material with possible booster injection, and follow-up of 12 months post injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Silk Microparticle Filler Injection (Experimental): A silk protein microparticle-based filler will be injected deep to the thyroarytenoid muscle of the paralyzed vocal fold to augment/medialize its position.
  Interventions: Procedure: Silk Microparticle Filler Injection

INTERVENTIONS:
Procedure: Silk Microparticle Filler Injection — A silk protein microparticle-based filler will be injected deep to the thyroarytenoid muscle of the paralyzed vocal fold to augment/medialize its position.

SUMMARY:
This study will investigate the safety and efficacy of a silk protein microparticle-based filler for vocal fold injection augmentation to treat dysphonia/dysphagia secondary to vocal fold paralysis. Participants will receive one injection and follow-up for a planned period of 12 months.

DETAILED DESCRIPTION:
Vocal fold paralysis is a clinical condition that arises commonly as a complication of surgery, endotracheal intubation, malignancy, or idiopathic etiologies. It often results in glottal insufficiency, which is the inability of the true vocal folds to meet and achieve complete closure during normal physiologic functions such as speech, swallowing, and coughing. The presence of vocal fold paralysis with glottal insufficiency can lead to decreased quality-of-life, as well as increase risks of complications such as aspiration pneumonia.

Current treatments for vocal fold paralysis are based around techniques to medialize the paralyzed vocal fold. One manner in which this is done is via injection of a filler or bulking agent into the vocal fold in order to augment it. Injection augmentation has many advantages including its minimally invasive nature, overall safety and low risk/complication rate, immediate clinical effect, and ability to perform it at the bedside or in-office. Various materials are used for injection augmentation including autologous fat, hyaluronic acid, collagen, carboxymethylcellulose, and calcium hydroxyapatite. However, all of the current injection choices have individual limitations such as temporary effect, unpredictability due to variable resorption by the body, unfavorable mechanical properties, and challenging handling attributes.

Silk is derived from the Bombyx mori silk worm and has a long history as a surgical biomaterial. Surgical scaffolds derived from silk have been used for reconstructive surgery, due to its ability to allow cellular infiltration and encourage tissue regeneration/remodeling. Given the potential advantages of such a material, Brown et al engineered and studied a novel silk protein microparticle-based filler material suitable for injection augmentation.

Patients with unilateral vocal fold paralysis identified at the study sites will be offered participation in this study to receive injection augmentation of the paralyzed vocal fold with the filler material under investigation. Outcome measures evaluated pre- and post-injection and over follow-up visits will include various patient reported quality of life indices, objective clinical assessments of voice, laryngeal videostroboscopy examinations, and acoustic/aerodynamic testing. The investigators hypothesize that the novel silk protein microparticle-based filler will have a favorable safety profile for use as an injectable material in the human larynx and it will produce durable clinical benefit lasting up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral vocal fold immobility with glottal insufficiency present for at least 2 weeks from onset
* Willingness to partake in study and follow-up as documented by signed informed consent

Exclusion Criteria:

* History of allergy/hypersensitivity to silk or silk containing products
* History of allergy/hypersensitivity to hyaluronic acid (HA) or HA containing products
* History of allergy/hypersensitivity to lidocaine or amide-based anesthetics
* History of an autoimmune condition
* Significant immunocompromised state (i.e. immunosuppression s/p transplantation)
* Pregnancy
* Active infection or inflammation in the larynx
* Comorbid known laryngeal conditions including but not limited to vocal fold scar, vocal tremor, laryngeal dystonia, etc. that would warrant other interventions for optimal treatment
* History of laryngeal surgery
* Life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by FDA/CBER Adverse Event Severity Grading Scale | 12 months
  Adverse event severity grading scale from 1 to 4, with grade 1 as mild, grade 2 as moderate, grade 3 as severe, and grade 4 potentially life-threatening.

SECONDARY OUTCOMES:
Quality of Life as assessed by Voice Handicap Index-10 (VHI-10) | 12 months
  VHI-10 is a patient questionnaire with 10 statements rated from 0 to 4 with overall scale 0-40.
Quality of Life as assessed by Vocal Fatigue Index (VFI) | 12 months
  VFI is a patient questionnaire with 19 statements rated from 0-4 with overall scale 0-76.
Quality of Life as assessed by Dyspnea Index (DI) | 12 months
  DI is a patient questionnaire with 10 statements rated from 0 to 4 with overall scale 0-40.
Quality of Life as assessed by Eating Assessment Tool (EAT-10) | 12 months
  EAT-10 is a patient questionnaire with 10 statements rated from 0 to 4 with overall scale 0-40.
Objective Vocal Quality as assessed by experts using the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) instrument | 12 months
  Blinded evaluations of audio voice recordings will be performed by laryngologists and speech-language pathologists using the CAPE-V, which grades overall severity, roughness, breathiness, strain, pitch, and loudness from 0-100.
Vocal Fold Appearance as assessed by experts using a modified version of the Voice-Vibratory Assessment with Laryngeal Imaging (VALI) form | 12 months
  Blinded assessments of recorded laryngeal videostroboscopy exams will be performed by laryngologists and speech-language pathologists using a modified version of the VALI, which is a graphical rating form to grade various components seen on stroboscopy.
Objective Acoustic Testing as assessed by fundamental frequency | 12 months
  Measurement of fundamental frequency (F0) during sustained vowel phonation.
Objective Acoustic Testing as assessed by Sound Pressure Level (SPL) | 12 months
  Measurement of minimum/maximum SPL during phonation.
Objective Acoustic Testing as assessed by Cepstral Peak Prominence (CPP) | 12 months
  Measurement of CPP during phonation.
Objective Aerodynamic Testing as assessed by Vital Capacity (VC) | 12 months
  Measurement of VC.
Objective Aerodynamic Testing as assessed by Maximum Phonation Time (MPT) | 12 months
  Measurement of MPT.
Objective Aerodynamic Testing as assessed by Mean Glottal Flow Rate (MGFR) | 12 months
  Measurement of MGFR.
Objective Aerodynamic Testing as assessed by Subglottal Pressure (SGP) | 12 months
  Measurement of SGP.
Objective Aerodynamic Testing as assessed by Cough Velocity (CV) | 12 months
  Measurement of maximum CV.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spector BC, Netterville JL, Billante C, Clary J, Reinisch L, Smith TL. Quality-of-life assessment in patients with unilateral vocal cord paralysis. Otolaryngol Head Neck Surg. 2001 Sep;125(3):176-82. doi: 10.1067/mhn.2001.117714. PMID 11555751
- [Background] Brown JE, Gulka CP, Giordano JEM, Montero MP, Hoang A, Carroll TL. Injectable Silk Protein Microparticle-based Fillers: A Novel Material for Potential Use in Glottic Insufficiency. J Voice. 2019 Sep;33(5):773-780. doi: 10.1016/j.jvoice.2018.01.017. Epub 2018 Mar 30. PMID 29609905
- [Background] Etienne O, Schneider A, Kluge JA, Bellemin-Laponnaz C, Polidori C, Leisk GG, Kaplan DL, Garlick JA, Egles C. Soft tissue augmentation using silk gels: an in vitro and in vivo study. J Periodontol. 2009 Nov;80(11):1852-8. doi: 10.1902/jop.2009.090231. PMID 19905955
- [Background] Bellas E, Panilaitis BJ, Glettig DL, Kirker-Head CA, Yoo JJ, Marra KG, Rubin JP, Kaplan DL. Sustained volume retention in vivo with adipocyte and lipoaspirate seeded silk scaffolds. Biomaterials. 2013 Apr;34(12):2960-8. doi: 10.1016/j.biomaterials.2013.01.058. Epub 2013 Jan 29. PMID 23374707
- [Background] Kijanska M, Marmaras A, Hegglin A, Kurtcuoglu V, Giovanoli P, Lindenblatt N. In vivo characterization of the integration and vascularization of a silk-derived surgical scaffold. J Plast Reconstr Aesthet Surg. 2016 Aug;69(8):1141-50. doi: 10.1016/j.bjps.2016.01.017. Epub 2016 Feb 5. PMID 26966076
- [Background] Rosen CA, Gartner-Schmidt J, Casiano R, Anderson TD, Johnson F, Remacle M, Sataloff RT, Abitbol J, Shaw G, Archer S, Zraick RI. Vocal fold augmentation with calcium hydroxylapatite: twelve-month report. Laryngoscope. 2009 May;119(5):1033-41. doi: 10.1002/lary.20126. PMID 19274731